CLINICAL TRIAL: NCT06165796
Title: The Effect of LASIK on the Calibration of IOL Formula Calculation: a Comparative Study
Status: Completed | Type: Observational
Sponsor: Taipei Nobel Eye Clinic (Other)
Responsible Party: Principal Investigator, Chao-Kai Chang, Dean, Taipei Nobel Eye Clinic
Other Study IDs: 004
Record Dates: First submitted 2023-12-04; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cataract Senile
MeSH Terms: interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- previous LASIK group
  Interventions: Device: routine cataract surgery and intraocular lens implantation
- previous non-LASIK group
  Interventions: Device: routine cataract surgery and intraocular lens implantation

INTERVENTIONS:
Device: routine cataract surgery and intraocular lens implantation — routine cataract surgery and intraocular lens implantation

SUMMARY:
Direct comparison study between previous LASIK or non-LASIK cataract eyes, the performance between non-LASIK and LASIK patients were (i) Ophthalmic examinations: UDVA, CDVA and uncorrected near visual acuity (UNVA) (40cm) and (ii) Refractive prediction error: defined as difference between postoperative sphere and target refraction.

ELIGIBILITY:
Inclusion Criteria:

* presence of cataract in both eyes
* corrected distance visual acuity under 20/40
* Phacoemulsification cataract surgery was arranged for both eyes

Exclusion Criteria:

* complicated cataract
* corneal opacities or irregularities
* corneal astigmatism > 1.50 diopter
* amblyopia, anisometropia
* surgical complications such as posterior capsular bag rupture or vitreous loss, IOL tilt or decentration
* coexisting ocular pathologies, glaucoma, non-dilating pupil, history of intraocular surgery, or retinopathy
* optic nerve or macular diseases
* refusal or unable to maintain follow-up.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clear corneal phacoemulsification and IOL implantation were performed by single surgeon Chao-Kai Chang. The surgical process involved topical anesthesia, a 3-step clear corneal incision (2.75 mm) at 180° (temporal in both eyes), a 5.0-mm continuous curvilinear capsulorhexis, phacoemulsification using the stop-and-chop technique, IOL implantation with an injector, IOL centration, and a sutureless incision. The study IOL models include only EDOF Symfony IOL (Johnson and Johnson, Santa Ana, CA, USA).
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | 1 month after surgery
refractive prediction error | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Nobel Eye Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abulafia A, Hill WE, Koch DD, Wang L, Barrett GD. Accuracy of the Barrett True-K formula for intraocular lens power prediction after laser in situ keratomileusis or photorefractive keratectomy for myopia. J Cataract Refract Surg. 2016 Mar;42(3):363-9. doi: 10.1016/j.jcrs.2015.11.039. Epub 2016 Mar 19. PMID 27006324
- [Result] Yeu E, Cuozzo S. Matching the Patient to the Intraocular Lens: Preoperative Considerations to Optimize Surgical Outcomes. Ophthalmology. 2021 Nov;128(11):e132-e141. doi: 10.1016/j.ophtha.2020.08.025. Epub 2020 Aug 31. PMID 32882308